CLINICAL TRIAL: NCT03628248
Title: Effect of Endovascular Inferior Mesenteric Artery Embolization on Colonic Perfusion Prior to Rectal Surgery for Rectal Tumor or Sigmoid Colon Surgery - A Single-center Feasibility Pilot Study.
Brief Title: Effect of Endovascular Inferior Mesenteric Artery Embolization on Colonic Perfusion Prior to Rectal Surgery for Rectal Tumor or Sigmoid Colon Surgery
Acronym: AMIREMBOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NIMAO/2017-02/JF-02; 2017-A03527-46 (Other: ANSM)
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2021-08

CONDITIONS: Cancer, Sigmoid; Cancer, Rectum
MeSH Terms: conditions — Sigmoid Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- embolization (Experimental)
  Interventions: Procedure: embolization of the inferior mesenteric artery; Procedure: Inferior mesenteric artery ligation
- No embolization (Other)
  Interventions: Procedure: Inferior mesenteric artery ligation

INTERVENTIONS:
Procedure: embolization of the inferior mesenteric artery — proximal occlusion of the inferior mesenteric artery, before its divisional branches, by coils or plug 3-4 weeks prior to surgery.
  Arms: embolization
Procedure: Inferior mesenteric artery ligation — Endovascular ligation of Inferior mesenteric artery

SUMMARY:
The investigators hypothesize that a primary embolization, 3-4 weeks before surgery, would allow development of vascular collaterality, in particular for the marginal artery which will ensure a better colonic perfusion.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is at least 18 years old and less than 80 years old
* Patient has rectal cancer or sigmoid colon cancer requiring surgical treatment

Exclusion Criteria:

* The subject is participating in another study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient has a history of abdominal surgery
* Patient suffers from a hemostasis disorder (hemophilia, von Willebrand disease, thrombocytopenia) and is on anticoagulant therapy.
* Patient whose general condition appears too precarious or is taking corticosteroids or immunosuppressants leading to an unacceptable surgical risk.
* Renal insufficiency with clearance <45ml / min
* Known allergy to contrast media
* Patient who had treatment of the abdominal aorta or its branches Reported pregnancy (the existence of effective contraception will be verified for women of childbearing age).
* Anatomical variant at risk or absence of marginal artery highlighted at the time of arteriography.
* Abnormality of the superior mesenteric artery
* Historic occlusion of the inferior mesenteric artery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-04-11 (Actual); Study Completion 2021-04-11 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation of the colon after inferior mesenteric artery ligation between groups | Prior to start of surgery
  Digital oxymeter (%)
Arterial pressure after inferior mesenteric artery ligation between groups | Prior to start of surgery
  Average (mmHg)
Colonic perfusion in the marginal artery after inferior mesenteric artery ligation between groups | Prior to start of surgery
  Rectal resistance index measured by Doppler
Oxygen saturation of the colon after inferior mesenteric artery ligation between groups | 60 seconds after surgery
  Digital oxymeter (%)
Oxygen saturation of the colon after inferior mesenteric artery ligation between groups | 5 minutes after surgery
  Digital oxymeter (%)
Arterial pressure in the marginal artery after inferior mesenteric artery ligation between groups | 60 seconds after surgery
  Average (mmHg)
Arterial pressure in the marginal artery after inferior mesenteric artery ligation between groups | 5 minutes after surgery
  Average (mmHg)
Colonic perfusion in the marginal artery after inferior mesenteric artery ligation between groups | 60 seconds after surgery
  Rectal resistance index measured by Doppler
Colonic perfusion in the marginal artery after inferior mesenteric artery ligation between groups | 5 minutes after surgery
  Rectal resistance index measured by Doppler

SECONDARY OUTCOMES:
Presence of post-embolization complications | Day 5 post-emoblization
  Yes/No
Presence of post-surgery complications | Hospital discharge (Day 7 after surgery)
  Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bertrand, MD, Principal Investigator — CHU Nimes
Locations (1):
- CHU Nimes, Nîmes, France

REFERENCES:
- [Result] Frandon J, Berny L, Prudhomme M, de Forges H, Serrand C, de Oliveira F, Beregi JP, Bertrand MM. Inferior mesenteric artery embolization ahead of rectal cancer surgery: AMIREMBOL pilot study. Br J Surg. 2022 Jul 15;109(8):650-652. doi: 10.1093/bjs/znac071. PMID 35333313